CLINICAL TRIAL: NCT07322510
Title: Health Behaviour Change, Education on Risk Factor Reduction, Physical Activity Guidance, and Nutrition Counselling With a Remote Team to Support Patient Progress Using Technology in Synchronization With Medication Management and CardioWatch 287-2. (HEARTS in Sync + CardioWatch 287-2)
Brief Title: HEARTS in Sync + CardioWatch 287-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Corsano Health B.V. (Industry)
Responsible Party: Principal Investigator, Nicholas Giacomantonio, Medical Director - REDUCE-IT, Cardiologist, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: REB File No. 1032019
Record Dates: First submitted 2025-11-18; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Wearable Device; Cardiovascular Disease; ASCVD Management; CHF - Congestive Heart Failure
Keywords: virtual cardiac rehabilitation; wearable device; remote monitoring
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Intervention Model Description: Participants enrolled in HEARTS in Sync program who use the Corsano CardioWatch 287-2 will be followed to evaluate the implementation and usability of the device into routine virtual cardiac rehabilitation care, as well as associated health outcomes. The health outcomes from participants in the clinical trial will be compared to two external control groups. First external control group consists of patients who are enrolled in usual care, virtual cardiac rehab program without the Corsano CardioWatch 287-2 device. The second external control group consists of patients who completed an on-site cardiac rehabilitation program. Both external control groups sign a program consent form that allows their data to be used for research purposes.
  This design allows for assessment of the device integration into usual care and its impact on patient outcomes in a real-world setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual Cardiac Rehab + Corsano CardioWatch 287-2 (Experimental)
  Interventions: Device: Remote Patient Monitoring with Corsano CardioWatch 287-2

INTERVENTIONS:
Device: Remote Patient Monitoring with Corsano CardioWatch 287-2 — Participants wear a CardioWatch 287-2 during the 13-week virtual cardiac rehabilitation program, HEARTS in Sync. The program is delivered by the Nova Scotia Health clinical team that consists of a Registered Nurse, Registered Dietitian and Physiotherapist.
  The CardioWatch 287-2 collects health information such as pulse rate, blood pressure, sleep, steps, activity, and more. This information is available for participants to check on the patient app called "Corsano". The information is also summarized on a weekly report that reports 7-day average which the clinical team will review on the Healthcare Practitioner web-based portal. This information is used to guide the participants rehabilitation journey.
  These participants will be followed to understand program adherence, patient-reported usability and acceptability, and clinical outcomes collected at baseline and program discharge.

SUMMARY:
The goal of this interventional study is to evaluate the implementation, usability, and clinical outcomes of a wearable medical-grade device in a virtual Cardiac Rehabilitation (CR) program, titled HEARTS in Sync. The question guiding this study is: Do patient clinical outcomes differ between those who use the CardioWatch 287-2 during the HEARTS in Sync program as compared to those who participate without using the CardioWatch 287-2? The comparison will happen between two non-randomized groups of patients who are enrolled in the HEARTS in Sync virtual CR program.

The wearable device (CardioWatch 287-2), worn on patient's wrists, will provide clinicians with physiological information to better mirror the clinical oversight provided to an in-person CR program. Participants who choose to use the device will be asked to wear it daily. The clinical team will review weekly summary reports to help guide participant progress through the 13-week program.

The primary objectives of this study are to:

1. Characterize participants (e.g., demographic health history, patient feedback) between those who choose to use the CardioWatch 287-2 device and those who do not.
2. Compare clinical outcomes between users and non-users of the device within the HEARTS in Sync program, by:

   1. Tracking patient enrollment, attendance in virtual education sessions, and program completion rates,
   2. Evaluating change in patient bloodwork outcomes,
   3. Measuring change is physical ability,
   4. Analyzing changes in eating behaviours, and
   5. Examining quality of life using validated tools.
3. Asses the feasibility of the CardioWatch 287-2 for the HEARTS in Sync virtual CR program by:

   1. Assessing device adherence
   2. Reviewing patient feedback survey, and
   3. Determining if clinician team were able to access and interpret data collected throughout the program

The secondary objective of this study is to compare clinical outcomes of device users during the HEARTS in Sync program with patients who completed the on-site CR program.

This research aims to better understand how a medical-grade device may improve virtual CR programming to extend clinical care to the community. As a result, this could lead to a more personalized care and better results for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet CR inclusion criteria requirements and who are enrolling in virtual cardiac rehab program, HEARTS in Sync, in Nova Scotia.

Exclusion Criteria:

Phones that are not compatible with the Corsano system.

* Huawei P8 Lite
* Huawei P9 Lite
* Xiaomi Mi 6
* Huawei P20 Lite
* Apple iOS version lower than 14.5
* Android OS version lower than 8.0
* Android or Apple devices without Bluetooth® 5.0 Low Energy capability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Patient Program Adherence | From enrollment to 13-week program completion
  The proportion (%) of program sessions attended by each patient, comparing device users and non-device user. Attendance percentage will be obtained by program records.
Change in Metabolic Equivalents (METs) from Baseline to Discharge Between Device Users and Non-Device Users | Baseline (after program assessment but before program start) and Discharge (near program completion, up to 6 weeks after program end)
  Change in Metabolic Equivalents measured during the baseline exercise stress test and discharge stress test.
Change in Fat Intake Score Between Device Users and Non-Device Users | Baseline (after program assessment but before program start) and Discharge (near program completion, up to 6 weeks after program end)
  Change in patient fat intake score measured using a validated nutrition questionnaire at baseline and discharge.
Change in Fibre Intake Score Between Device Users and Non-Device Users | Baseline (after program assessment but before program start) and Discharge (near program completion, up to 6 weeks after program end)
  Change in patient fibre intake score measured using a validated nutrition questionnaire at baseline and discharge.
Change in Sodium Intake Score Between Device Users and Non-Device Users | Baseline (after program assessment but before program start) and Discharge (near program completion, up to 6 weeks after program end)
  Change in patient sodium intake score measured using a validated nutrition questionnaire at baseline and discharge.
Change in Sugar Intake Score Between Device Users and Non-Device Users | Baseline (after program assessment but before program start) and Discharge (near program completion, up to 6 weeks after program end)
  Change in patient fat intake score measured using a validated nutrition questionnaire at baseline and discharge.
Change in Quality of Life Ladder Score Between Device Users and Non-Device Users | Baseline (after program assessment but before program start) and Discharge (near program completion, up to 6 weeks after program end)
  Examine change in patient-reported quality of life using the Quality of Life Ladder at initial/baseline and discharge report.
Change in Satisfaction with Life Between Device Users and Non-Device Users | Baseline (after program assessment but before program start) and Discharge (near program completion, up to 6 weeks after program end)
  Examine change in patient-reported quality of life using the Satisfaction with Life Scale at initial/baseline and discharge report.
Characterize Participants | Initial (at assessment)
  Determine demographic and health history between device users and non-device users
Device Adherence to Wearing the CardioWatch 287-2 | From enrollment to the end of the program at 13-weeks
  Device adherence will be assessed by calculating the proportion of total study days during which each participant wore the device for the required monitoring duration. Adherence will be categorized into one of the three following groups:
  1. High compliance: ≥ 50% daily wear time (~12 hours/day on all 7 days/week)
  2. Moderate compliance: ≥ 25% daily wear time (~6 hours/day)
  3. Low compliance: ≥ 12.5% daily wear time (~3 hours/day)
  The unit of measure is percentage (%) of days with required wear time and proportion (%) of participants in each adherence category.
  Device adherence is automatically captured through the Corsano CardioWatch 287-2 system.
Patient-Reported Usability and Acceptability of the CardioWatch 287-2 | After completion of the program (e.g. after 13 weeks)
  Participants' perceptions of usability, comfort, and acceptability of the device will be assessed using a study-specific questionnaire that includes both participant rating scale and free-text responses. Only the ranked items will be used for quantitative outcome reporting while the free-text responses will be summarized descriptively.
Clinician-Reported Usability of the CardioWatch 287-2 System | Up to 1 year after study completion
  Clinicians' assessment of device usability including ease of data interpretation, integration into clinical workflow, and perceived clinical value. This will be a descriptive analysis only captured through a study-specific focus group.
Change in Triglyceride Level Change Between Device Users and Non-Device Users | Baseline (after assessment but before program start) and Discharge (near end of program or up to 6 weeks after program completion)
  Triglycerides (mmol/L) will be measured via standard blood panel.
Change in Total Cholesterol Level Change Between Device Users and Non-Device Users | Baseline (after assessment but before program start) and Discharge (near end of program or up to 6 weeks after program completion)
  Total cholesterol (mmol/L) will be measured via lipid panel in bloodwork.
Change in HDL Cholesterol Level Change Between Device Users and Non-Device Users | Baseline (after assessment but before program start) and Discharge (near end of program or up to 6 weeks after program completion)
  HDL cholesterol (mmol/L) will be measured via lipid panel in bloodwork.
Change in LDL Cholesterol Level Change Between Device Users and Non-Device Users | Baseline (after assessment but before program start) and Discharge (near end of program or up to 6 weeks after program completion)
  LDL cholesterol (mmol/L) will be measured via lipid panel in bloodwork.
Change in Hemoglobin A1C Level Change Between Device Users and Non-Device Users | Baseline (after assessment but before program start) and Discharge (near end of program or up to 6 weeks after program completion)
  HbA1C (%) will be measured via standard bloodwork.
Change in Systolic Blood Pressure Between Device Users and Non-Device Users | Baseline (between assessment and program start) and Discharge (near end of program or up to 6 weeks after program completion)
  Systolic blood pressure (mmHg) measured by a blood pressure monitor.
Change in Diastolic Blood Pressure Between Device Users and Non-Device Users | Baseline (between assessment and program start) and Discharge (near end of program or up to 6 weeks after program completion)
  Diastolic blood pressure (mmHg) measured by a blood pressure monitor.
Change in Resting Heart Rate between Device Users and Non-Device Users | Initial (at assessment) and Discharge (near end of program completion, up to 6 weeks after program completion)
  Resting heart rate (beats per minute) will be measured at assessment and near end of program completion

SECONDARY OUTCOMES:
Change in Metabolic Equivalents (METs) from Baseline to Discharge Between Device Users and In-Person Patients | Baseline (after assessment but before program start) and Discharge (near end of program or up to 6 weeks after program completion)
  Change in Metabolic Equivalents measured during the baseline exercise stress test and discharge stress test.
Change in Fat Intake Score Between Device Users and In-Person Patients | Baseline (after program assessment but before program start) and Discharge (near program completion, up to 6 weeks after program end)
  Change in patient fat intake score measured using a validated nutrition questionnaire at baseline and discharge.
Change in Fibre Intake Score Between Device Users and In-Person Patients | Baseline (after program assessment but before program start) and Discharge (near program completion, up to 6 weeks after program end)
  Change in patient fibre intake score measured using a validated nutrition questionnaire at baseline and discharge.
Change in Sodium Intake Score Between Device Users and In-Person Patients | Baseline (after program assessment but before program start) and Discharge (near program completion, up to 6 weeks after program end)
  Change in patient sodium intake score measured using a validated nutrition questionnaire at baseline and discharge.
Change in Sugar Intake Score Between Device Users and In-Person Patients | Baseline (after program assessment but before program start) and Discharge (near program completion, up to 6 weeks after program end)
  Change in patient fat intake score measured using a validated nutrition questionnaire at baseline and discharge.
Change in Quality of Life Ladder Score Between Device Users and In-Person Patients | Baseline (after program assessment but before program start) and Discharge (near program completion, up to 6 weeks after program end)
  Examine change in patient-reported quality of life using the Quality of Life Ladder at initial/baseline and discharge report.
Change in Satisfaction with Life Between Device Users and In-Person Patients | Baseline (after program assessment but before program start) and Discharge (near program completion, up to 6 weeks after program end)
  Examine change in patient-reported quality of life using the Satisfaction with Life Scale at initial/baseline and discharge report.
Change in Triglyceride Level Change Between Device Users and In-Person Patients | Baseline (after assessment but before program start) and Discharge (near end of program or up to 6 weeks after program completion)
  Triglycerides (mmol/L) will be measured via standard blood panel.
Change in Total Cholesterol Level Change Between Device Users and In-Person Patients | Baseline (after assessment but before program start) and Discharge (near end of program or up to 6 weeks after program completion)
  Total cholesterol (mmol/L) will be measured via lipid panel in bloodwork.
Change in HDL Cholesterol Level Change Between Device Users and In-Person Patients | Baseline (after assessment but before program start) and Discharge (near end of program or up to 6 weeks after program completion)
  HDL cholesterol (mmol/L) will be measured via lipid panel in bloodwork.
Change in LDL Cholesterol Level Change Between Device Users and In-Person Patients | Baseline (after assessment but before program start) and Discharge (near end of program or up to 6 weeks after program completion)
  LDL cholesterol (mmol/L) will be measured via lipid panel in bloodwork.
Change in Hemoglobin A1C Level Change Between Device Users and In-Person Patients | Baseline (after assessment but before program start) and Discharge (near end of program or up to 6 weeks after program completion)
  HbA1C (%) will be measured via standard bloodwork.
Change in Systolic Blood Pressure Between Device Users and In-Person Patients | Baseline (between assessment and program start) and Discharge (near end of program or up to 6 weeks after program completion)
  Systolic blood pressure (mmHg) measured by a blood pressure monitor.
Change in Diastolic Blood Pressure Between Device Users and In-Person Patients | Baseline (between assessment and program start) and Discharge (near end of program or up to 6 weeks after program completion)
  Diastolic blood pressure (mmHg) measured by a blood pressure monitor.
Change in Resting Heart Rate between Device Users and In-Person Patients | Initial (at assessment) and Discharge (near end of program completion, up to 6 weeks after program completion)
  Resting heart rate (beats per minute) will be measured at assessment and near end of program completion

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas B Giacomantonio, Medical Doctor, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Mumford Professional Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corsano Health BV. CardioWatch 287-2 Bracelet & Mobile Patient App Instruction Manual.; 2024. www.corsano.com
- [Background] van Vliet M, Monnink SHJ, Kuiper MJ, Constandse JC, Hoftijzer D, Ronner E. Evaluation of a novel cuffless photoplethysmography-based wristband for measuring blood pressure according to the regulatory standards. Eur Heart J Digit Health. 2024 Feb 8;5(3):335-343. doi: 10.1093/ehjdh/ztae006. eCollection 2024 May. PMID 38774367
- [Background] Blok S, Piek MA, Tulevski II, Somsen GA, Winter MM. The accuracy of heartbeat detection using photoplethysmography technology in cardiac patients. J Electrocardiol. 2021 Jul-Aug;67:148-157. doi: 10.1016/j.jelectrocard.2021.06.009. Epub 2021 Jul 2. PMID 34256184
- [Background] Monnink SHJ, van Vliet M, Kuiper MJ, Constandse JC, Hoftijzer D, Muller M, Ronner E. Clinical evaluation of a smart wristband for monitoring oxygen saturation, pulse rate, and respiratory rate. J Clin Monit Comput. 2025 Apr;39(2):451-457. doi: 10.1007/s10877-024-01229-z. Epub 2024 Oct 10. PMID 39388061
- [Background] Stas P. Corsano Health Receives EU-MDR Certification. https://corsano.com/corsano-health-receives-eu-mdr-certification/.
- [Background] Verhaar C. Corsano Health Receives FDA Clearance. https://corsano.com/28091-2/.
- [Background] van Deudekom T. Corsano Health Receives ISO 13485 Certification. https://corsano.com/medical-certification/.
- [Background] Jones AK, Yan CL, Rivera Rodriquez BP, Kaur S, Andrade-Bucknor S. Role of wearable devices in cardiac telerehabilitation: A scoping review. PLoS One. 2023 May 31;18(5):e0285801. doi: 10.1371/journal.pone.0285801. eCollection 2023. PMID 37256878
- [Background] Yeghiazarians Y, Jneid H, Tietjens JR, Redline S, Brown DL, El-Sherif N, Mehra R, Bozkurt B, Ndumele CE, Somers VK. Obstructive Sleep Apnea and Cardiovascular Disease: A Scientific Statement From the American Heart Association. Circulation. 2021 Jul 20;144(3):e56-e67. doi: 10.1161/CIR.0000000000000988. Epub 2021 Jun 21. PMID 34148375
- [Background] Cheung C. The Emerging Role of Wearables in Cardiac Care. Vol 100.; 2023.
- [Background] Pare G, Leaver C, Bourget C. Diffusion of the Digital Health Self-Tracking Movement in Canada: Results of a National Survey. J Med Internet Res. 2018 May 2;20(5):e177. doi: 10.2196/jmir.9388. PMID 29720359
- [Background] Bayoumy K, Gaber M, Elshafeey A, Mhaimeed O, Dineen EH, Marvel FA, Martin SS, Muse ED, Turakhia MP, Tarakji KG, Elshazly MB. Smart wearable devices in cardiovascular care: where we are and how to move forward. Nat Rev Cardiol. 2021 Aug;18(8):581-599. doi: 10.1038/s41569-021-00522-7. Epub 2021 Mar 4. PMID 33664502
- [Background] Lear SA. The Delivery of Cardiac Rehabilitation Using Communications Technologies: The "Virtual" Cardiac Rehabilitation Program. Can J Cardiol. 2018 Oct;34(10 Suppl 2):S278-S283. doi: 10.1016/j.cjca.2018.07.009. Epub 2018 Jul 18. PMID 30274638
- [Background] Lam J, Ahmad K, Gin K, Chow CM. Deliver Cardiac Virtual Care: A Primer for Cardiovascular Professionals in Canada. CJC Open. 2022 Feb;4(2):148-157. doi: 10.1016/j.cjco.2021.10.001. Epub 2021 Oct 9. PMID 34661090
- [Background] Ramachandran HJ, Jiang Y, Tam WWS, Yeo TJ, Wang W. Effectiveness of home-based cardiac telerehabilitation as an alternative to Phase 2 cardiac rehabilitation of coronary heart disease: a systematic review and meta-analysis. Eur J Prev Cardiol. 2022 May 25;29(7):1017-1043. doi: 10.1093/eurjpc/zwab106. PMID 34254118
- [Background] Moulson N, Bewick D, Selway T, Harris J, Suskin N, Oh P, Coutinho T, Singh G, Chow CM, Clarke B, Cowan S, Fordyce CB, Fournier A, Gin K, Gupta A, Hardiman S, Jackson S, Lamarche Y, Lau B, Legare JF, Leong-Poi H, Mansour S, Marelli A, Quraishi AUR, Roifman I, Ruel M, Sapp J, Small G, Turgeon R, Wood DA, Zieroth S, Virani S, Krahn AD. Cardiac Rehabilitation During the COVID-19 Era: Guidance on Implementing Virtual Care. Can J Cardiol. 2020 Aug;36(8):1317-1321. doi: 10.1016/j.cjca.2020.06.006. Epub 2020 Jun 14. PMID 32553606
- [Background] Dalal HM, Doherty P, McDonagh ST, Paul K, Taylor RS. Virtual and in-person cardiac rehabilitation. BMJ. 2021 Jun 3;373:n1270. doi: 10.1136/bmj.n1270. No abstract available. PMID 34083376
- [Background] Thomas RJ, Beatty AL, Beckie TM, Brewer LC, Brown TM, Forman DE, Franklin BA, Keteyian SJ, Kitzman DW, Regensteiner JG, Sanderson BK, Whooley MA. Home-Based Cardiac Rehabilitation: A Scientific Statement From the American Association of Cardiovascular and Pulmonary Rehabilitation, the American Heart Association, and the American College of Cardiology. J Am Coll Cardiol. 2019 Jul 9;74(1):133-153. doi: 10.1016/j.jacc.2019.03.008. Epub 2019 May 13. PMID 31097258
- [Background] Brouwers RWM, van Exel HJ, van Hal JMC, Jorstad HT, de Kluiver EP, Kraaijenhagen RA, Kuijpers PMJC, van der Linde MR, Spee RF, Sunamura M, Uszko-Lencer NHMK, Vromen T, Wittekoek ME, Kemps HMC; Committee for Cardiovascular Prevention and Cardiac Rehabilitation of the Netherlands Society of Cardiology. Cardiac telerehabilitation as an alternative to centre-based cardiac rehabilitation. Neth Heart J. 2020 Sep;28(9):443-451. doi: 10.1007/s12471-020-01432-y. PMID 32495296
- [Background] Scherrenberg M, Wilhelm M, Hansen D, Voller H, Cornelissen V, Frederix I, Kemps H, Dendale P. The future is now: a call for action for cardiac telerehabilitation in the COVID-19 pandemic from the secondary prevention and rehabilitation section of the European Association of Preventive Cardiology. Eur J Prev Cardiol. 2021 May 14;28(5):524-540. doi: 10.1177/2047487320939671. PMID 32615796
- [Background] Santiago de Araujo Pio C, Beckie TM, Varnfield M, Sarrafzadegan N, Babu AS, Baidya S, Buckley J, Chen SY, Gagliardi A, Heine M, Khiong JS, Mola A, Radi B, Supervia M, Trani MR, Abreu A, Sawdon JA, Moffatt PD, Grace SL. Promoting patient utilization of outpatient cardiac rehabilitation: A joint International Council and Canadian Association of Cardiovascular Prevention and Rehabilitation position statement. Int J Cardiol. 2020 Jan 1;298:1-7. doi: 10.1016/j.ijcard.2019.06.064. Epub 2019 Jul 4. PMID 31405584
- [Background] Grace SL, Bennett S, Ardern CI, Clark AM. Cardiac rehabilitation series: Canada. Prog Cardiovasc Dis. 2014 Mar-Apr;56(5):530-5. doi: 10.1016/j.pcad.2013.09.010. Epub 2013 Oct 11. PMID 24607018
- [Background] Owen O, O'Carroll V. The effectiveness of cardiac telerehabilitation in comparison to centre-based cardiac rehabilitation programmes: A literature review. J Telemed Telecare. 2024 May;30(4):631-646. doi: 10.1177/1357633X221085865. Epub 2022 Apr 4. PMID 35369770
- [Background] Grace SL, Turk-Adawi K, Santiago de Araujo Pio C, Alter DA. Ensuring Cardiac Rehabilitation Access for the Majority of Those in Need: A Call to Action for Canada. Can J Cardiol. 2016 Oct;32(10 Suppl 2):S358-S364. doi: 10.1016/j.cjca.2016.07.001. Epub 2016 Jul 9. PMID 27692116
- [Background] Jamal Z, Horn R, Ager A. Effect of contributing factors on the incidence of non-communicable diseases among adults with common mental health disorders: a systematic review [Internet]. Southampton (UK): National Institute for Health and Care Research; 2024 May 22. Available from http://www.ncbi.nlm.nih.gov/books/NBK612376/ PMID 40014738
- [Background] Dalal HM, Doherty P, Taylor RS. Cardiac rehabilitation. BMJ. 2015 Sep 29;351:h5000. doi: 10.1136/bmj.h5000. No abstract available. PMID 26419744
- [Background] Mizuno A, Changolkar S, Patel MS. Wearable Devices to Monitor and Reduce the Risk of Cardiovascular Disease: Evidence and Opportunities. Annu Rev Med. 2021 Jan 27;72:459-471. doi: 10.1146/annurev-med-050919-031534. Epub 2020 Sep 4. PMID 32886543